CLINICAL TRIAL: NCT06438211
Title: Comparison of Postoperative Analgesic Effectiveness of Superficial and Deep Serratus Plane Blocks in Patients Undergoing Mastectomy
Brief Title: Comparison of Postoperative Analgesic Effectiveness of Superficial and Deep Serratus Plane Blocks for Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ayse Ulgey, Professor doctor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024/58
Record Dates: First submitted 2024-05-09; First posted 2024-05-31 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2024-05

CONDITIONS: Mastectomy; Postoperative Pain; Analgesia
Keywords: serratus anterior plane block; local anesthetic; regional anesthesia; postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Mastectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (superficial serratus anterior plane block) (Active Comparator): Single-shot ultrasound (Esaote Mylab30) guided Superficial SAP block with 30 ml 0.25% bupivacain (Marcain 0.5%, Astra Zeneca, Turkey) at the T4- T5 ribs level (between the latissimus dorsi muscle and the serratus anterior muscle) was performed preoperatively to patients in the Superficial SAP group (Group I)
  Interventions: Procedure: superficial or deep serratus anterior plane block for mastectomy
- Group II (deep serratus anterior plane block) (Active Comparator): Single- shot ultrasound (Esaote Mylab30) guided Deep SAP block with 30 ml 0.25% bupivacain (Marcain 0.5%, Astra Zeneca, Turkey) at the T4- T5 ribs level ( between the serratus anterior muscle and the ribs) was performed preoperatively to patients in the Deep SAP group (Group I)
  Interventions: Procedure: superficial or deep serratus anterior plane block for mastectomy

INTERVENTIONS:
Procedure: superficial or deep serratus anterior plane block for mastectomy — group I: superficial SAP Block for postoperative analgesia for mastectomy group II: deep SAP Block for postoperative analgesia for mastectomy

SUMMARY:
Pain after breast surgery can be quite severe and can significantly affect quality of life. By successfully treating acute pain, it is aimed to prevent the formation of pain memory and to ensure that chronic pain never occurs. It is known that by using regional techniques, the use of general anesthetics and opioids can be reduced and their harmful effects can be limited. In this study, it will be compared the analgesic effectiveness of superficial and deep serratus plane blocks in the postoperative acute and chronic periods.

DETAILED DESCRIPTION:
Acute and chronic pain is a serious problem in patients undergoing breast surgery. Apart from the feeling of pain, it also causes psychological difficulties, increased hospital stays, delays or difficulties in mobilization, and so on. Due to all these reasons, postoperative pain control is very important.

Although opioids are the gold standard in the treatment of pain, their side effect profiles (sedation, respiratory depression, constipation, tolerance development, etc.) limit their use and different searches are on the agenda. There are studies showing that superficial and deep serratus plane blocks are effective in mastectomy operations. In this study, patients who underwent mastectomy these two blocks will be compared to see which one is superior and to investigate the differences that may occur in the acute and chronic periods.

After general anesthesia induction, a superficial serratus plane block will be performed on the first group of patients undergoing surgery by applying local anesthetic to the fascia between the serratus anterior and latissimus dorsi muscles at the level of the 4th and 5th ribs under ultrasound. then the patient will undergo surgical procedure. Likewise, for the second group of patients, after general anesthesia induction, a deep serratus plane block will be performed by applying local anesthetic between the rib and the serratus anterior muscle at the level of the 4th and 5th ribs, under ultrasound guidance, and the patient will be taken into surgery. Both groups of patients will be monitored for 24 hours after the operation with a patient-controlled analgesia device. Patients' pain scores, satisfaction scores, nausea and vomiting scores, and additional analgesic needs will be recorded 24 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* patients who will undergo mastectomy surgery
* patients who agreed to participate in the study
* ASA I-II patients

Exclusion Criteria:

* Patients planned for bilateral breast surgery
* Patients who have had previous breast surgery
* Patients with existing neuropathic pain or receiving treatment for neuropathic pain
* Patients with psychiatric disorders
* Patients with opioid addiction
* Patients allergic to local anesthetics

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Since breast cancer is much more common in women than men and to ensure homogenization in the study, only female patients will be included.
Enrollment: 63 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
postoperative morphine consumption | 24 hours
  How much morphine the patient consumed in the first 24 hours postoperatively with a patient-controlled anesthesia device

SECONDARY OUTCOMES:
measuring pain scors | 24 hours
  Determining patients' pain levels with a visual analog scale (VAS) between the scale of 1-10

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Ülgey, MD, Study Director — TC Erciyes University
Locations (1):
- University of Erciyes, Kayseri, Talas, Turkey (Türkiye)